CLINICAL TRIAL: NCT04620265
Title: Differential Air Pressure Technology for Improving Gait Performance and Reducing Fall Risk in Diabetic Elderly Saudi Patients
Brief Title: Differential Air Pressure Technology for Treatment of Diabetic Elderly Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Shamekh Mohamed El-Shamy, Professor, Umm Al-Qura University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: Umm AlQura Univ
Record Dates: First submitted 2020-10-31; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-03

CONDITIONS: Diabetic Polyneuropathy
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Weight-Bearing

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Treadmill training 100% (Experimental): This group received antigravity treadmill training 100% weight bearing and conventional exercise program.
  Interventions: Other: Antigravity treadmill training 100% weight bearing; Other: The conventional exercise program
- Treadmill training 75% (Experimental): This group received antigravity treadmill training 75% weight bearing and conventional exercise program.
  Interventions: Other: Antigravity treadmill training 75% weight bearing; Other: The conventional exercise program
- Treadmill training 50% (Experimental): This group received antigravity treadmill training 50% weight bearing and conventional exercise program.
  Interventions: Other: Antigravity treadmill training 50% weight bearing; Other: The conventional exercise program
- Treadmill training 25% (Experimental): This group received antigravity treadmill training 25% weight bearing and conventional exercise program.
  Interventions: Other: Antigravity treadmill training 25% weight bearing; Other: The conventional exercise program
- Conventional program (Sham Comparator): This group received the conventional exercise program only.
  Interventions: Other: The conventional exercise program

INTERVENTIONS:
Other: Antigravity treadmill training 100% weight bearing — This group received antigravity treadmill training 100% weight bearing and conventional exercise program.
  Arms: Treadmill training 100%
Other: Antigravity treadmill training 75% weight bearing — This group received antigravity treadmill training 75% weight bearing and conventional exercise program.
  Arms: Treadmill training 75%
Other: Antigravity treadmill training 50% weight bearing — This group received antigravity treadmill training 50% weight bearing and conventional exercise program.
  Arms: Treadmill training 50%
Other: Antigravity treadmill training 25% weight bearing — This group received antigravity treadmill training 25% weight bearing and conventional exercise program.
  Arms: Treadmill training 25%
Other: The conventional exercise program — This group received the conventional exercise program only.

SUMMARY:
Aging can be defined as sequential deterioration that occurs in elderly people including weakness, loss of mobility, decline of physical capabilities, increase susceptibility to disease and many other age-related physiological changes .The beginning of old age in most developed countries is about 60 or 65 years old. Diabetes mellitus (DM) and most commonly type 2 DM is one of the most common chronic non-communicable diseases affecting old people in Saudi Arabia which might be resulted from decline in physical activities. Polyneuropathy (PN) and its serious consequences represent the most common complication in diabetic mellitus which could contribute to an increased gait abnormality and risk of falling.

DETAILED DESCRIPTION:
Disability and reduction of quality of life are the largest costs of diabetes and its complications. So taking active intervention to reduce the risk of falls, improve gait performance and improve the quality of life in elderly with DPN is very important. Lower extremity aerobic exercise training via treadmill aiming for improving patients' physical activity levels is an important part in the rehabilitation program to enhance balance and walking functions and reducing the fall risk, .Treadmill training using s low-load walking provided by an emerging technology called lower body positive pressure (LBPP) that effectively reduces body weight could be preferable than other methods of unweighting treadmill because the air pressure is applied uniformly over the lower body. This kind of anti-gravity treadmill is ideal in reducing the formation of pain and pressure points that are common with harness-based unweighting systems. Many other advantages are also associated with this unique type of antigravity technology that could give it the superiority than the other types of unweighting treadmills in enhancing walking performance, reducing the risk of fall and improving quality of life in Saudi elderly people with DPN.

ELIGIBILITY:
Inclusion Criteria:

* Elderly Saudi men with diabetic polyneuropathy with history of 2 or more falls within the past 12 months
* Diagnosed as having uncontrolled Type 2 Diabetes Mellitus, with glycosylated haemoglobin (HbA1c) level between 7 and 11 and fasting glucose level ranged from 7.0 -11.1 mmol/L.
* Treated only with oral anti-diabetic agents (not taking insulin),
* Pharmacological treatment had to be stable for at least 3 months before the study.
* They will be selected among old subjects that were able to walk independently with or without assistive device but with poor balance

Exclusion Criteria:

* Type 1 Diabetes Mellitus,
* Patients who had got a score over 19 according to Tinetti scale of balance assessment,
* Patient with malnutrition (BMI < 21 kg/m2 or with recent weight loss > 5% body weight in the last month or > 10% in six months),
* Patients with established hypertension (resting systolic blood pressure > 140 mmHg and diastolic blood pressure > 90 mmHg,
* With any severe chronic or uncontrolled comorbid condition as recent myocardial infarction, unstable angina, acute congestive heart failure, third degree heart block and uncontrolled arrhythmia.
* Patients will be excluded also if they have abnormal skin integrity e.g. wound or scare tissues or are on other complementary treatment,
* History of serious cerebrovascular or cardiovascular diseases, and severe debilitating musculoskeletal problems).

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline functional capacity at 3 months | Baseline and 3 months post-intervention
  The assessment of functional capacity will be done using Six Minute Walk Test where intensity is moderately higher than daily living activities. Subject will be asked to walk at his own maximal pace from end to end of a 40-meter flat, straight corridor marked every 1 meter with side cones, in order to cover as much ground as possible while maintaining a steady pace without running during the allowed time. No verbal encouragement will be given, and subjects will be informed verbally each 2 minutes of the remaining time. The patients will be allowed to stop, but they can start again, if possible, within the allocated 6 minutes. Distance covered in 6 minutes will be recorded in meter. The longer the distance that will be walked will signify a better performance.
Change from baseline Health Related Quality of Life at 3 months | Baseline and 3 months post-intervention
  For assessment of Health Related Quality of Life, 36-item Medical Outcomes Study Short Form Questionnaire (Arabic version) will be used. Dimensions are physical functioning, social functioning, bodily pain, limitations caused by physical health problems; limitations caused by emotional problems, emotional well-being and mental health, energy-fatigue and vitality, general health perception. Participants' scores for Questionnaire will be computed following the protocol of Ware and associates and the higher scores mean better outcome.
Change from baseline Mobility at 3 months | Baseline and 3 months post-intervention
  Assessment of Mobility using Tinetti Performance Oriented Mobility Assessment. This is a widely recognized objective instrument for determining balance and gait deficiencies and assessing the risk of future falls. Higher Tinetti scores (maximum 28) correlate inversely with risk of falls. Individuals with Tinetti scores under 19 are considered to be at the highest risk for falls, those with scores between 19 and 24 are considered to have a moderate risk of falling, and those with scores 24 and above are considered to be at low risk for falls.
Change from baseline fall risk at 3 months | Baseline and 3 months post-intervention
  Fall risk assessment by using Balance Biodex stability system
Change from baseline spatial and temporal gait parameters at 3 months | Baseline and 3 months post-intervention
  Gait parameters assessment by using the GAITRite system. The main measured parameters will be step and stride length (cm), step width (cm), step time (sec), stance to swing ratio (%), cadence (steps/min) and velocity cm/sec.

CONTACTS AND LOCATIONS:
Overall Officials: Shamekh M El-Shamy, Ph.D., Principal Investigator — Professor
Locations (1):
- Al Noor Specialized Hospital, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No